CLINICAL TRIAL: NCT02847910
Title: ClinicaI Observation of Induced Abortion With Disposable Tissue Suction Tube
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014KTCC 03-05
Record Dates: First submitted 2016-06-05; First posted 2016-07-28 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Early Pregnancy
Keywords: tissue suction tube; disposable instrument; induced abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): device： High-tech disposable tissue suction set for uterine cavity tissue is produced by Xi'an Mejiajia Medical Equipment Company ; The participants will be use the disposable tissue suction set during the induced abortion procedure.
  Interventions: Procedure: the disposable tissue suction set
- control group (Experimental): device： Traditional metal instruments for induced abortion procedure; The participants will be use traditional metal instruments during induced abortion procedure.
  Interventions: Procedure: traditional metal instruments of abortion

INTERVENTIONS:
Procedure: the disposable tissue suction set — Induced abortion is a main backstop for terminating unwanted pregnancies, however, traditional hard metal instruments has lots of insufficiencies such as easily tissue damage, and repeatedly sterilization increases the incidence of cross infection in the hospital what leads to more complications of pelvic inflammation, infertility and so on. Therefore disposable non-metallic instruments are desperately needed as a way to decrease the complications and provide better medical services to patients. So, the investigators want to explore the clinical effect of disposable tissue suction tube set and make comparison with traditional metal instruments.
  Arms: experimental group
Procedure: traditional metal instruments of abortion — Induced abortion is a main backstop for terminating unwanted pregnancies. In Chinese hospital, traditional metal instruments are always used during the surgery. So the investigators want to explore the clinical effect of disposable tissue suction tube set and make comparison with traditional metal instruments.
  Arms: control group

SUMMARY:
The purpose of this study is to explore the clinical effect of disposable tissue suction tube set for induced abortion and make comparison with traditional metal instruments．

ELIGIBILITY:
Inclusion Criteria:

* premedical abortion diagnosed by ultrasound diagnosed
* pregnancy for the first time
* 7-9 weeks of pregnancy
* voluntary termination of pregnancy
* without surgical contraindication

Exclusion Criteria:

* refuse this clinical trial
* with systemic disease such as hypertensive disease, heart disease, diabetes
* refuse to terminate the pregnancy

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
blood loss (ml) | up to 5-10 minutes
  It always takes 5-10 minutes to finish the induced abortion in the outpatient, so the investigators will measure the blood loss during the operation time.
the rate of induced abortion syndrome (%); | up to 5-10 minutes
  It always takes 5-10 minutes to finish the induced abortion in the outpatient, so the investigators will observe whether induced abortion syndrome happens to our patients during the operation time.

SECONDARY OUTCOMES:
evaluate pain grade (0, I, II, III) by questionnaire | up to 5-10 minutes
  The participants will be asked some questions on questionnaire about feeling to evaluate their pain grade.
rate of leaving bed in 5 min by patient self (%) | 5 min after the surgery
operation time (minutes) | up to 5-10 minutes until the operation finished
  measure the operation time
the success rate of induced abortion (%) | up to 15 days after the surgery
  Ultrasound and gynecological examinations will be used to calculate the success rate of induced abortion.

CONTACTS AND LOCATIONS:
Overall Officials: Qiling Li, MD, PHD, Principal Investigator — The First Affliated Hospital of Xi'an Jiaotong University
Locations (1):
- The First Affliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juarez F, Singh S. Incidence of induced abortion by age and state, Mexico, 2009: new estimates using a modified methodology. Int Perspect Sex Reprod Health. 2012 Jun;38(2):58-67. doi: 10.1363/3805812. PMID 22832146
- [Background] Vilela RC, Benchimol M. Trichomonas vaginalis and Tritrichomonas foetus: interaction with fibroblasts and muscle cells - new insights into parasite-mediated host cell cytotoxicity. Mem Inst Oswaldo Cruz. 2012 Sep;107(6):720-7. doi: 10.1590/s0074-02762012000600003. PMID 22990959
- [Background] Albers CE, Steppacher SD, Ganz R, Siebenrock KA, Tannast M. Joint-preserving surgery improves pain, range of motion, and abductor strength after Legg-Calve-Perthes disease. Clin Orthop Relat Res. 2012 Sep;470(9):2450-61. doi: 10.1007/s11999-012-2345-0. PMID 22528379